CLINICAL TRIAL: NCT06944665
Title: The Palliative Effect of TENS-WAA on 'Capsaicin/Heat' Induced Acute Lower Back Pain: a Self-controlled Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaonan Huang (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Huang, researcher, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Organization: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHEC2025-005
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Acute Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left (Experimental): At the time of the first phase of the trial: analgesic intervention in the left lower ankle after capsaicin/heat pain modelling in the left subject area adjacent to the 2nd-4th lumbar vertebrae in the Left1 group of subjects.At the time of the second phase of the trial: analgesic intervention in the left lower ankle after capsaicin/heat pain modelling in the right subject area adjacent to the 2nd-4th lumbar vertebrae in the Left group of subjects.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory
- Right (Experimental): At the time of the first phase of the trial: subjects in the Right1 group underwent analgesic intervention in the right lower ankle after capsaicin/heat pain modelling in the right subject area adjacent to the 2nd-4th lumbar vertebrae.At the time of the second phase of the trial: subjects in the Right1 group underwent analgesic intervention in the right lower ankle after capsaicin/heat pain modelling in the left subject area adjacent to the 2nd-4th lumbar vertebrae.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory — Based on the theory of wrist and ankle needles, transcutaneous electrical nerve stimulation is a kind of analgesic treatment device that combines wrist and ankle needles with transcutaneous electrical nerve stimulation, and can be worn on the human wrist and ankle. Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture Theory uses low-frequency electronic pulses to stimulate the entry point of the wrist-ankle needle, which has the advantages of easy to wear, concentration of the treatment site, safety of the treatment, and no needles.

SUMMARY:
Acute lower back pain is a common condition that occurs in all age groups, and most people will experience acute lower back pain at least once in their lives. The use of pharmacological analgesic interventions may result in complications such as gastrointestinal reactions, skin reactions, and renal damage, so there is an urgent need for an analgesic method that is easy to use, relatively safe, and has no significant systemic side effects to alleviate patients' pain.

Wrist and ankle acupuncture is an acupuncture therapy developed by Professor Zhang Xinshu and other professors of the First Affiliated Hospital of the Second Military Medical University of the Chinese People's Liberation Army based on the meridian theory of Chinese medicine, by dividing the human body into two segments and six zones and treating them according to the longitudinal zones in which the illnesses are located or the corresponding points of the areas where the primary lesions are located, in order to achieve the purpose of dredging the meridians and collaterals, regulating qi and blood, balancing the yin and yang, relieving pain and treating the illnesses, and it has been widely used for treating the clinical It is widely used to treat all kinds of pain and neurological diseases.

Transcutaneous Electrical Nerve Stimulation is a non-invasive pain treatment method, which relieves pain by distributing current of specific frequency and intensity to stimulate peripheral nerves. In recent years, our team has combined the wrist and ankle needles with transcutaneous electrical nerve stimulation to develop an analgesic device that can be worn on the human wrist and ankle, which is called transcutaneous electrical nerve stimulation based on the theory of wrist and ankle needles. Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory（TENS-WAA) uses low-frequency electronic pulses to stimulate the entry point of the wrist-ankle acupuncture needle, which has the advantages of easy to wear, concentrated treatment site, safe treatment, and needle-free.

Functional near-infrared spectroscopy is a novel optical technique for non-invasive brain activity measurement by reading cerebral haemodynamics and oxygen saturation. Advantages include portability, non-invasiveness, no ionising radiation or drug injections, and simultaneous measurement of two haemodynamic parameters - deoxyhaemoglobin and oxyhaemoglobin. Several studies have demonstrated the utility and potential of functional NIR spectroscopy for pain assessment.

In medical research, the capsaicin model is widely used to simulate acute pain in humans, and capsaicin-induced pain sensations are produced primarily through binding to capsaicin receptors. Topical application of capsaicin activates TRPV1, located at the end of primary sensory neurons in the trunk and viscera, which, through a series of actions, leads to the release of pro-inflammatory factors, while injury receptors in the skin then generate neural signals that are transferred to the cerebral cortex, resulting in the sensation of pain. The sensation is similar to neuropathic pain, and pro-inflammatory factors also play a key role in the pathophysiological process of acute lower back pain. Therefore, the use of capsaicin is effective in inducing acute lower back pain, while related studies have shown that the combination of heat and capsaicin has a synergistic or additive effect.

The present study was designed as an autocross-control study in which a 'capsaicin-thermal pain' low back model was established in healthy subjects to induce acute lower back pain, and the analgesic efficacy of TENS-WAA was verified by using the fNIRS, VAS, and other assessment methods, with the following main objectives:

1. To repeat the validity of the pre-cortical fNIRS pain assessment paradigm in a controlled study;
2. To validate the efficacy of the Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory intervention in an autocross-control study by using fNIRS to collect data on changes in blood oxygen levels in brain regions involved in pain perception (frontal pole area and dorsolateral prefrontal cortex), as well as the VAS;
3. Explore the specificity of Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory acupoints through the self-randomised crossover control of 'unilateral pain + ipsilateral intervention' and 'unilateral pain + contralateral intervention'.

DETAILED DESCRIPTION:
Content of the study Phase 1 trial: subjects were randomly divided into Left1 group (n=15) and Right1 group (n=15), subjects in the Left1 group were intervened in the left lower ankle after capsaicin/heat pain modelling in the left region adjacent to the lumbar vertebrae of L2-L4; subjects in the Right1 group were intervened in the right lower ankle after capsaicin/heat pain modelling in the right region adjacent to the lumbar vertebrae of L2-L4. Intervention.

Phase 2 trial: subjects in the Left1 and Right1 groups of the Phase 1 trial were crossed over, i.e., the Left1 group was assigned to the Right2 group and the Right1 group was assigned to the Left2 group. the Left2 group intervened in the right lower ankle after capsaicin/heat pain modelling was established in the left region adjacent to the lumbar vertebrae of L2-L4, and the Right2 group intervened in the right lower ankle in the right region adjacent to the lumbar vertebrae of L2-L4. After establishing the capsaicin/heat pain model, the intervention was performed on the left lower ankle.

Research Methods

1. Experimental environment A quiet, dark and undisturbed indoor environment was selected, with a constant room temperature of 26°C, and the subjects were kept in a sitting position throughout the experiment to facilitate the acquisition of functional near infrared spectroscopy (fNIRS) signals.
2. Test materials Functional near infrared spectroscopy (fNIRS) signal acquisition equipment, transcutaneous electrical nerve stimulation equipment based on the theory of carpal and ankle needling, capsaicin cream (CAPZASIN-HP, 0.1% capsaicin), medical alcohol disinfectant wet wipes, cling film, and temperature-controlled hot packs.
3. Capsaicin sensitivity test Capsaicin sensitivity test was first performed on the included subjects by applying capsaicin cream on the inner left forearm of the subjects 1cm×1cm, with a thickness of about 1mm. retaining the capsaicin for 5min, and subjects with allergic reactions and capsaicin intolerance were excluded from the test.
4. Lower back capsaicin-heat pain model In this experiment, the capsaicin-thermal pain model was established by applying hot compresses with capsaicin cream: capsaicin cream (CAPZASIN-HP, 0.1% capsaicin) was applied to two symmetrical areas of 5 cm × 10 cm on either side of the alcohol sterilised lumbar paraspinal region of L2-L4, at a thickness of approximately 2 mm, and covered with cling film, and a hot compress bag with a constant temperature of 40°C was used to apply hot compresses on the area for for 10 minutes, and the application position was as shown in Figure 1. Capsaicin was retained throughout and wiped off at the end of the trial.
5. Methods Using an own-crossover controlled study, subjects (n=30) included in the trial were subjected to two phases of the trial, separated by a washout period of more than 7 days. Before the start of the trial, the subjects were educated about the trial process and pain assessment methods. The transcutaneous electrical nerve stimulation (TENS-WAA) action site based on the theory of wrist and ankle acupuncture (TENS-WAA) was selected from the lower 5 or 6 sites on the lateral side of the ankle according to the records of Practical Wrist and Ankle Acupuncture and literature references, which can treat low back pain, lumbar spine and paravertebral pain, and sciatica.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males between the ages of 18-44 years;
* The dominant hand is the right hand;
* No persistent pain in the last month;
* No acute pain in the last week;
* Good health with no medical condition for which he/she is receiving treatment;
* Subjects agreed to participate in this trial and signed an informed consent form.

Exclusion Criteria:

* With malignant tumours and serious heart, liver and kidney diseases;
* Those with skin breakage at the site of capsaicin application;
* Those with a history of lumbar spine surgery, spinal fracture, rheumatic disease, cancer, pacemaker, or congenital anomalies of the spine;
* Any other medical condition that may affect pain perception, including neurological and psychiatric disorders;
* Taking sedative and sleep-aiding drugs within one week;
* Those who are allergic to capsaicin;
* Currently participating in another clinical trial concerning lower back pain or pain.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
functional near-infrared spectroscopy | Throughout the entire experimental procedure (up to 50 minutes)

SECONDARY OUTCOMES:
Short-Form McGill Pain Questionnaire | at 10 minutes post capsaicin/heat-induced pain modeling ,at 10 minutes post electrical stimulation ,at 20 minutes post electrical stimulation
  The Simplified McGill Pain Questionnaire includes three items: The first is the Pain Rating Index (PRI), which encompasses 11 sensory descriptors and 4 affective descriptors. Each term is scored on a scale of 0-3 based on pain intensity, with a maximum score of 45 and a minimum of 0 (higher scores indicate greater pain).
  The second item is the Visual Analog Scale (VAS), primarily consisting of a 10 cm line where 0 represents "no pain at all" and 10 signifies "the worst pain imaginable," with higher scores indicating greater pain.
  The third item is the Present Pain Intensity (PPI), categorized into 6 levels: 0 = no pain, 1 = mild, 2 = discomforting, 3 = distressing, 4 = horrible, 5 = excruciating.
Oxygen | Throughout the entire experimental procedure (up to 50 minutes)
heart rate | Throughout the entire experimental procedure (up to 50 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China